CLINICAL TRIAL: NCT07236723
Title: Vitamin D, Nerve Growth Factor and Nerve Conduction Studies in Adult Male Type 2 Diabetic Neuropathy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Marwa Nasry Elbadry, Instructor of medical physiology, Aswan University
Other Study IDs: diabetic neuropathy
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Neuropathy
Keywords: vitamin d, nerve growth factor and diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Hereditary Sensory and Autonomic Neuropathies | interventions — Nerve Growth Factor; Vitamin D

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: Group І: Control group included non-diabetic healthy males aged (40-60) years old
  Interventions: Other: 25(OH) vitamin D
- type 2 diabetic male not suffering from diabetic neuropathy aged(40-60) years old: type 2 diabetic male not suffering from diabetic neuropathy aged(40-60) years old
  Interventions: Other: Nerve Growth Factor
- type2 diabetic males suffering from diabetic neuropathy aged(40_60)years old: type2 diabetic males suffering from diabetic neuropathy aged(40_60)years old
  Interventions: Other: nerve conduction studies

INTERVENTIONS:
Other: nerve conduction studies — Assessment of neuropathy by nerve conduction studies of sural and tibial nerves in both lower extremities.
  Groups: type2 diabetic males suffering from diabetic neuropathy aged(40_60)years old
Other: Nerve Growth Factor — nerve growth factor level using its corresponding ELISA kit
  Groups: type 2 diabetic male not suffering from diabetic neuropathy aged(40-60) years old
Other: 25(OH) vitamin D — 25(OH) vitamin D serum level using its corresponding ELISA kit
  Groups: control group

SUMMARY:
study the relationship of vitamin d with nerve growth factor level and nerve conduction studies in adult male type 2 diabetic neuropathy patients

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) is one of the most frequent microvascular complications of both type1 (T1DM) and type2 diabetes mellitus (T2DM) . It involves damage to the peripheral nerves, leading to symptoms such as numbness, tingling, pain, and loss of sensation in the extremities, especially the feet and hands . It is the primary risk factor for lower limb ulcers, amputations and consequent disabling, that can significantly affect a person's quality of life.

Unfortunately, the exact pathogenesis of diabetic neuropathy is complex and multifactorial. However, several studies have shown that increased levels of blood glucose leads to several neuronal changes as accumulation of advanced glycation end products, mitochondrial impairment and DNA damage. Furthermore, Vitamin D deficiency is more common in people with T2DM, contributing its pathogenesis in many ways, including impairment of insulin secretion and increasing insulin resistance. Moreover, previous studies reported that low level of vitamin D is correlated with the presence and severity of sensory neuropathy . However, its pathogenesis has not yet been established.

Nerve growth factor (NGF) is a neurotrophic factor playing a major role in adult peripheral nerve system. It works by increasing nerve cell regeneration and decreasing degeneration, so NGF decreased levels induce peripheral nerve lesion in diabetic patients.

Several studies indicate that vitamin D may play a role in nutrition and protection of peripheral nerves as nerve cells and glial cells rich in vitamin D receptors, So vitamin D may have a potential effect in DPN by neuro-protection as it protect against apoptosis and degeneration, as well as it can trigger production of NGF helping preservation of neurons. Thus, we hypothesize that vitamin D, by regulating NGF expression, could help nerve regeneration and improve outcomes in patients with DPN.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients 40 -65 years' old who have type 2 diabetes mellitus on oral hypoglycemic , non-diabetic healthy subjects of matched age and type 2male diabetic neuropathy patients of matched age .

Exclusion Criteria:

* Cardiac patients.
* Patients who have transient ischemic attack or stroke.
* Patients with inflammatory rheumatic diseases.
* Patients with malignant diseases.
* Hyperparathyroidism.
* Hypothyroidism.
* Renal impairment with renal replacement therapy.
* Liver diseases.
* Patients on vitamin D supplementation.
* Patients on vitamin B12 supplementation.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group І: Control group included non-diabetic healthy males. Group П: Type 2 male diabetic patients not suffering from diabetic neuropathy in Aswan University Hospital of matched age.
  Group III: Type 2 male diabetic patients suffering from diabetic neuropathy in Aswan University Hospital of matched age.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
study the relation of vitamin d and nerve growth factor with nerve conduction studies in type 2 diabetic neuropathy male patients | one year
  1. Difference in vitamin D level between diabetic neuropathy patients, diabetic patients without neuropathy and healthy subjects.
  2. Difference in serum nerve growth factor level between diabetic neuropathy patients, diabetic patients without neuropathy and healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan university hospital, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
no need

REFERENCES:
- [Result] Shafiee A, Rafiei MA, Jafarabady K, Eskandari A, Abhari FS, Sattari MA, Amini MJ, Bakhtiyari M. Effect of cannabis use on blood levels of brain-derived neurotrophic factor (BDNF) and nerve growth factor (NGF): A systematic review and meta-analysis. Brain Behav. 2024 Jan;14(1):e3340. doi: 10.1002/brb3.3340. PMID 38376038
- [Result] Pittas AG, Jorde R, Kawahara T, Dawson-Hughes B. Vitamin D Supplementation for Prevention of Type 2 Diabetes Mellitus: To D or Not to D? J Clin Endocrinol Metab. 2020 Dec 1;105(12):3721-33. doi: 10.1210/clinem/dgaa594. PMID 32844212
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC7571449/
- Available data/document: Data Monitoring Committee Charter — https://pmc.ncbi.nlm.nih.gov/articles/PMC7571449/ — https://pmc.ncbi.nlm.nih.gov/articles/PMC7571449/